CLINICAL TRIAL: NCT06035497
Title: A Phase 1/2 Study of the Safety, Tolerability, Pharmacokinetics, and Efficacy of BMS-986369 (Golcadomide) in Participants With Relapsed or Refractory T-cell Lymphomas in Japan (GOLSEEK-3)
Brief Title: A Study to Assess the Safety, Tolerability, Efficacy, and Drug Levels of BMS-986369 (Golcadomide) in Participants With Relapsed or Refractory T-cell Lymphomas in Japan (GOLSEEK-3)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA073-1008
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Relapsed or Refractory T-cell Lymphomas
Keywords: Relapsed or Refractory Peripheral T-cell Lymphoma (R/R PTCL); Relapsed or Refractory Adult T-cell Leukemia/Lymphoma (R/R ATL); Golcadomide; BMS-986369; CC-99282; Adult T-cell leukemia/lymphoma (ATL); Peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS); Angioimmunoblastic T-cell lymphoma and other nodal lymphomas of T follicular helper (TFH) cell origin; Angioimmunoblastic T-cell lymphoma (AITL); Follicular T-cell lymphoma (FTCL); Nodal peripheral T-cell lymphoma with TFH phenotype; Anaplastic large cell lymphoma, ALK-positive (ALCL, ALK+); Anaplastic large cell lymphoma, ALK-negative (ALCL, ALK-); Breast implant-associated anaplastic large cell lymphoma (BIA-ALCL); Extranodal NK/T-cell lymphoma, nasal type (ENKL); Mycosis fungoides (MF)
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell; Lymphoma, T-Cell, Peripheral; Leukemia-Lymphoma, Adult T-Cell; Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Extranodal NK-T-Cell; Mycosis Fungoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Administration of BMS-986369 (Experimental)
  Interventions: Drug: BMS-986369

INTERVENTIONS:
Drug: BMS-986369 — Specified dose on specified days
  Other Names: Golcadomide; CC-99282

SUMMARY:
The purpose of this study is to test the safety, tolerability, efficacy, and drug levels of BMS-986369 (Golcadomide) in participants with relapsed or refractory T-cell lymphomas in Japan (GOLSEEK-3).

ELIGIBILITY:
Inclusion Criteria

- Have one of the following subtypes of T-cell Lymphoma (TCL) with relapsed or refractory disease, as assessed by the investigator:.

i) Adult T-cell leukemia-lymphoma (ATL).

ii) Peripheral T-cell lymphoma not otherwise specified (PTCL-NOS).

iii) Angioimmunoblastic T-cell lymphoma (AITL) and other nodal lymphomas of T follicular helper phenotype (TFH) cell origin.

iv) Anaplastic large cell lymphoma (ALCL), anaplastic lymphoma kinase-positive (ALK+).

v) ALCL, anaplastic lymphoma kinase-negative (ALK-).

vi) Breast implant-associated ALCL.

vii) Extranodal NK/T-cell lymphoma, nasal type (ENKL).

viii) Mycosis fungoides (MF) with advanced stage (stage IIB-IVB).

* Phase 1 participants must not be responsive, intolerant, or ineligible to standard therapies that may prolong life or provide symptomatic relief, or for whom no standard therapeutic option is available in the clinical practice guidelines in the opinion of the investigator.
* Phase 2 participants must have been treated by at least 1 prior line of systemic therapy.
* Have an Eastern Cooperative Oncology Group performance status of 0, 1 or 2.

Exclusion Criteria

* Have any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participants from participating in the study.
* Have any condition, including active or uncontrolled infection, or the presence of laboratory abnormalities, which places the participants at unacceptable risk if he/she were to participate in the study.
* Have a life expectancy ≤ 3 months.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2030-10-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 5 weeks after last dose of treatment
  Phase 1 participants
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 5 weeks after last dose of treatment
  Phase 1 participants
Number of participants with Dose-Limiting Toxicity (DLT) | Up to 28 days after first dose
  Phase 1 participants
Number of participants with laboratory abnormalities | Up to 5 weeks after last dose of treatment
  Phase 1 participants
Number of participants with vital sign abnormalities | Up to 5 weeks after last dose of treatment
  Phase 1 participants
Number of participants with Electrocardiogram (ECG) abnormalities | Up to 5 weeks after last dose of treatment
  Phase 1 participants
Eastern Cooperative Oncology Group Performance Status (ECOG PS) | Up to 5 weeks after last dose of treatment
  Phase 1 participants
Number of participants with Left Ventricular Ejection Fraction (LVEF) assessment abnormalities | Up to 5 weeks after last dose of treatment
  Phase 1 participants
Number of participants with Physical Examination (PE) abnormalities | Up to 5 weeks after last dose of treatment
  Phase 1 participants
Number of participants who achieve Objective Response (OR) as assessed by central review per international consensus response criteria for ATL | Up to 2 years after last does of treatment
  Phase 2: Adult T-cell Leukemia-Lymphoma (ATL) cohort
  OR is defined as the achievement of Partial Response (PR), complete response unconfirmed (CRu), or Complete Response (CR)
Number of participants who achieve OR as assessed by central review per protocol-defined response criteria according to Lugano classification (Computed Tomography(CT)-based) | Up to 2 years after last dose of treatment
  Phase 2: Peripheral T-cell Lymphoma (PTCL) cohort
  OR is defined as the achievement of PR or CR

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 8 of Cycle 2 (each cycle is 28 days)
Area under the plasma concentration time-curve (AUC) | Up to Day 8 of Cycle 2 (each cycle is 28 days)
Time to peak (maximum) plasma concentration (Tmax) | Up to Day 8 of Cycle 2 (each cycle is 28 days)
Number of participants with AEs | Up to 5 weeks after last dose of treatment
  Phase 2 participants
Number of participants with TEAEs | Up to 5 weeks after last dose of treatment
  Phase 2 participants
Number of participants with laboratory abnormalities | Up to 5 weeks after last dose of treatment
  Phase 2 participants
Number of participants with vital sign abnormalities | Up to 5 weeks after last dose of treatment
  Phase 2 participants
Number of participants with ECG abnormalities | Up to 5 weeks after last dose of treatment
  Phase 2 participants
ECOG PS | Up to 5 weeks after last dose of treatment
  Phase 2 participants
Number of participants with LVEF assessment abnormalities | Up to 5 weeks after last dose of treatment
  Phase 2 participants
Number of participants with PE abnormalities | Up to 5 weeks after last dose of treatment
  Phase 2 participants
Number of participants who achieve OR as assessed by central review per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL participants
  OR is defined as the achievement of PR, CRu, or CR
Number of participants who achieve OR as assessed by investigator per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL participants
  OR is defined as the achievement of PR, CRu, or CR
Number of participants who achieve OR as assessed by central review per protocol defined response criteria according to Lugano classification (CT-based). | Up to 4 years after last dose of treatment
  PTCL participants
  OR is defined as the achievement of PR or CR
Number of participants who achieve OR as assessed by investigator per protocol defined response criteria according to Lugano classification (CT-based). | Up to 4 years after last dose of treatment
  PTCL participants
  OR is defined as the achievement of PR or CR
Number of participants who achieve disease control as assessed by central review per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL participants
  Disease control is considered to be stable disease (SD), PR, CRu, or CR
Number of participants who achieve disease control as assessed by investigator per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL participants
  Disease control is considered to be SD, PR, CRu, or CR
Number of participants who achieve CR as assessed by central review per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL participants
Number of participants who achieve CR as assessed by investigator per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL participants
Time to response (TTR) as assessed by central review per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL participants
TTR as assessed by investigator per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL participants
Duration of response (DOR) as assessed by central review per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL Participants
DOR as assessed by investigator per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL Participants
Progression Free Survival (PFS) as assessed by central review per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL participants
PFS as assessed by investigator per international consensus response criteria for ATL | Up to 4 years after last dose of treatment
  ATL participants
Number of participants who achieve disease control as assessed by central review per protocol defined response criteria according to Lugano classification (CT-based) | Up to 4 years after last dose of treatment
  PTCL participants
  Disease control is considered to be SD, PR or CR
Number of participants who achieve disease control as assessed by investigator per protocol defined response criteria according to Lugano classification (CT-based) | Up to 4 years after last dose of treatment
  PTCL participants
  Disease control is considered to be SD, PR or CR
Number of participants who achieve CR as assessed by central review per protocol defined response criteria according to Lugano classification (CT-based) | Up to 4 years after last dose of treatment
  PTCL participants
Number of participants who achieve CR as assessed by investigator per protocol defined response criteria according to Lugano classification (CT-based) | Up to 4 years after last dose of treatment
  PTCL participants
TTR as assessed by central review per protocol defined response criteria according to Lugano classification (CT-based) | Up to 4 years after last dose of treatment
  PTCL participants
TTR as assessed by investigator per protocol defined response criteria according to Lugano classification (CT-based) | Up to 4 years after last dose of treatment
  PTCL participants
DOR as assessed by central review per protocol defined response criteria according to Lugano classification (CT-based) | Up to 4 years after last dose of treatment
  PTCL participants
DOR as assessed by investigator per protocol defined response criteria according to Lugano classification (CT-based) | Up to 4 years after last dose of treatment
  PTCL participants
PFS as assessed by central review per protocol defined response criteria according to Lugano classification (CT-based) | Up to 4 years after last dose of treatment
  PTCL participants
PFS as assessed by investigator per protocol defined response criteria according to Lugano classification (CT-based) | Up to 4 years after last dose of treatment
  PTCL participants
Time to next treatment (TTNT) | From the date of last dose until the date of death, lost to follow-up, withdrawal of consent from the entire study, time to next treatment or the end of the trial, whichever occurs first, assessed up to 2 years after end of treatment.
Overall survival (OS) | From the date of last dose until the date of death, lost to follow-up, withdrawal of consent from the entire study, or the end of the trial, whichever occurs first, assessed up to 2 years after end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bistol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (40):
- Japan (40):
  - Anjo Kosei Hospital, Anjo-shi, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Kameda General Hospital, Kamogawa, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - International University of Health and Welfare Narita Hospital, Narita, Chiba
  - Aso Iizuka Hospital, Iizuka, Fukuoka
  - Japan Community Healthcare Organization Kyushu Hospital, Kitakyushu-shi, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Tokai University Hospital, Isehara, Kanagawa
  - Yokosukakyosai, Yokosuka, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - National Hospital Organization Nagasaki Medical Center, Ōmura, Nagasaki
  - Sasebo City General Hospital, Sasebo, Nagasaki
  - Kindai University Hospital- Osakasayama Campus, Ōsaka-sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashiku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Imamura General Hospital, Kagoshima
  - Kagoshima University Hospital, Kagoshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Kumamoto University, Kumamoto
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Kyorin University Hospital, Mitaka
  - University of Miyazaki Hospital, Miyazaki
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Okayama University Hospital, Okayama
  - Nakagami Hospital Okinawa, Okinawa
  - Osaka International Cancer Institute, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Oita Prefectural Hospital, Ōita

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html